CLINICAL TRIAL: NCT07166887
Title: Pharmacokinetics, Pharmacological Effects and Safety of Multi Dose of 7.5mg Tolvaptan Tablet in Healthy Male Subjects
Brief Title: Phase I Study Multi Dose of 7.5mg Tolvaptan in Health Male
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-11-808-01
Record Dates: First submitted 2025-08-22; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 7.5mg Tolvaptan multi dosing group (Experimental)
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — One dose on the first day and one dose on days 3-9, for a total of eight doses.

SUMMARY:
pharmacokinetics, pharmacological effects and safety of multi dose of 7.5mg Tolvaptan tablet in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Male, sign informed consent;
2. When signing the informed consent, the age range is 18-40 years old (including the upper and lower limits);
3. The body weight is not less than 50kg, and the body mass index is in the range of 19 ~ 24 (including the upper and lower limits);
4. According to the results of medical history, serological examination (HIV antibody, HBsAg, HCV antibody and syphilis antibody), physical examination, vital signs (temperature, blood pressure, pulse), 12-lead electrocardiogram, laboratory examination (blood routine, blood biochemistry, coagulation function and urine routine), etc., the subjects are certified as healthy.

Exclusion Criteria:

1. Patients with a history of heart, liver, kidney, digestive tract, metabolic, respiratory, blood, mental, nervous system and other disorders, and doctors judge that they are not suitable.
2. Patients with a history of various types of arrhythmias judged by the researchers to have clinical significance, including a history of familial genetic disease (a history of arrhythmias with a genetic tendency in relatives), and a history of rapid and slow arrhythmias, such as atrioventricular transmission Conduction block, sinus arrest, supraventricular tachycardia and so on.
3. Have a history, allergy or tendency to drugs and any other substances.
4. Known intolerance to components of the test drug, including lactose. For example, people with rare genetic galactose intolerance, lactase deficiency, or glucose-galactose malabsorption.
5. Various voiding disorders (frequent urination, or difficulty urinating, etc.).
6. People who smoke, drink or depend on other drugs.
7. Blood donors had an equivalent amount of blood loss (>350 ml) during the 12 weeks prior to enrollment.
8. Participated in any drug trials within 12 weeks prior to enrollment.
9. People who have taken preventive or therapeutic drugs in the last 2 weeks.
10. Consumed grapefruit or foods containing grapefruit in the week prior to administration.
11. In the investigator's judgment, the subject's diet deviates significantly from the normal intake of protein, carbohydrates, and fats (for example, vegetarian or vegan).
12. Have a history of postural hypotension (refers to a blood pressure drop of ≥20/10mmHg when the blood pressure changes from the lying position to the standing position, accompanied by dizziness and other symptoms), standing vertigo, collapse, syncopation, and vertigo.
13. Quiet for more than 3 minutes, sitting resting pulse below 55 beats/min or more than 90 beats/min.
14. Quiet for more than 3 minutes, sitting systolic blood pressure is lower than 100mmHg or higher than 140mmHg; Or diastolic depression of 60mmHg or more than 90mmHg.
15. Clinically significant 12-lead electrocardiogram abnormalities.
16. Clinically significant abnormalities in physical examination.
17. Positive for any of the serological tests for HIV antibodies, HBsAg, HCV antibodies and syphilis antibodies.
18. Other circumstances that the investigator determines may affect the subject's completion of the test.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06-07 (Actual); Primary Completion 2011-07-27 (Actual); Study Completion 2011-07-27 (Actual)

PRIMARY OUTCOMES:
Tolvaptan Pharmacokinetic | - On Day 1: 0.5 hour before the first dose - the Day 9th pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, day 24 (only on Day 2 and Day 10th morning), 36 ( on Day 2 and Day 10th everning) and 48 hours - Day 4th to 8th day pre-dose
  peak concentration (Cmax)
Tolvaptan Pharmacokinetic | On Day 1: 0.5 hour before the first dose - the Day 9th pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, day 24 (only on Day 2 and Day 10th morning), 36 ( on Day 2 and Day 10th everning) and 48 hours - Day 4th to 8th day pre-dose
  time to peak (Tmax)
Tolvaptan Pharmacokinetic | On Day 1: 0.5 hour before the first dose - the Day 9th pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, day 24 (only on Day 2 and Day 10th morning), 36 ( on Day 2 and Day 10th everning) and 48 hours - Day 4th to 8th day pre-dose
  area under the drug-time curve (AUC0-t and AUC0-∞)
Tolvaptan Pharmacokinetic | On Day 1: 0.5 hour before the first dose - the Day 9th pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, day 24 (only on Day 2 and Day 10th morning), 36 ( on Day 2 and Day 10th everning) and 48 hours - Day 4th to 8th day pre-dose
  elimination half-life (t1/2)
Tolvaptan Pharmacokinetic | On Day 1: 0.5 hour before the first dose - the Day 9th pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, day 24 (only on Day 2 and Day 10th morning), 36 ( on Day 2 and Day 10th everning) and 48 hours - Day 4th to 8th day pre-dose
  apparent clearance (CL/F)
Tolvaptan Pharmacokinetic | On Day 1: 0.5 hour before the first dose - the Day 9th pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, day 24 (only on Day 2 and Day 10th morning), 36 ( on Day 2 and Day 10th everning) and 48 hours - Day 4th to 8th day pre-dose
  apparent volume of distribution (Vd/F)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Liu H, Liu T, Liu M, Zheng X, Zhong W, Zhao Q, Jiang J, Hu P, Li Y. Clinical trial on the pharmacokinetics, pharmacodynamics and safety of tolvaptan in healthy Chinese males: an open-label, single and multiple dosage, parallel group study. Front Pharmacol. 2025 Nov 21;16:1713702. doi: 10.3389/fphar.2025.1713702. eCollection 2025. PMID 41357896